CLINICAL TRIAL: NCT03145545
Title: Expanded Access Protocol Using TCR Alpha/Beta T Cell/CD19+ Depleted Donor Peripheral Stem Cells
Brief Title: Expanded Access Protocol Using Alpha/Beta T and CD19+ Depleted PBSC
Status: Available | Type: Expanded Access
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Timothy Olson, Medical Director, Hematopoietic Stem Cell Transplantation (HSCT) Program, Children's Hospital of Philadelphia
Other Study IDs: 16-013527
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Leukemia; Bone Marrow Failure Syndrome; Immunodeficiencies
MeSH Terms: conditions — Leukemia; Bone Marrow Failure Disorders; Immunologic Deficiency Syndromes

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Device: Apha/beta T and CD19+ cell depletion using CliniMACS device — Stem cells will be processed using the CliniMACS device for alpha/beta and CD19+ T cell depletion. Processing of cells using the CliniMACS will occur in accordance with the Investigator Brochure and Technical Manual following the laboratory standard operating procedures (SOPs) and using aseptic technique.

SUMMARY:
The primary objective of this protocol is to expand access for patients who lack a fully HLA (Human leukocyte antigen) matched sibling donor, and who are candidates for allogeneic hematopoietic stem cell transplant (HSCT). These patients have a serious or immediately life-threatening disease for which HSCT is indicated. These patients are not eligible for other Children's Hospital of Philadelphia Institutional Review Board (IRB) approved protocols that utilize CliniMACs technology for T depletion.

DETAILED DESCRIPTION:
Only 25-30% of patients who may benefit from HSCT have a matched related donor. An unrelated cord blood may not be available due to size or matching criteria, or if a reduced intensity regiment is recommended. The risk of severe graft vs. host disease (GVHD) and other complications is higher with unrelated donors, or partially matched related donors. At the Children's Hospital of Philadelphia (CHOP) there is extensive experience using mismatched unrelated donors or partially matched related donors with complete or partial T depletion to reduce the risk of severe GVHD.

ELIGIBILITY:
PATIENT AND DONOR ELIGIBILITY

Patients who lack an HLA matched sibling and who are candidates for allogeneic hematopoietic stem cell transplant (HSCT) but do not meet criteria for current open institutional protocols using CliniMACs device for β T/CD19+ depletion. Patients with matched related donors including matched sibling donors may also be eligible if special clinical indications are met.

Patients with the following transplantable diseases:

Non-malignant diseases:

* Metabolic storage diseases correctable by HSCT
* Bone marrow failure syndromes
* Immunodeficiencies/immune dysregulation syndromes
* Sickle cell disease or thalassemia
* Other diseases treated with HSCT

Malignant diseases:

* Acute leukemias
* Chronic leukemias
* Lymphomas
* Myelodyplastic syndrome

Patient Eligibility criteria:

It is important to note that the conditioning prescribed to the patient will be determined based on the disease and organ status and will include agents that are standard. Appropriate combinations of chemotherapy, immunotherapy and/or radiation will be determined on an individual basis.

Patient eligibility will be assessed as per our institutional standard operating procedures:

* Signed informed consent
* Lansky or Karnofsky performance ≥ 60
* Hematologic and Organ Function as per current institutional SOP
* Infectious Evaluation as per current institutional SOP
* Participants of childbearing potential must have a negative pregnancy test as per institutional SOP
* Subjects with graft failure who require a second HSCT will not need to meet eligibility criteria again prior to the second transplant. Graft failure is a medical emergency that requires HSCT

Donor Eligibility Patients must have an identified living donor

* Donor selection will comply with 21 CFR 1271*
* Unrelated donor that meets the matching criteria of the NMDP with allele matching at HLA -A, -B, -C, -DRB1, and -DQB1: Unrelated donors may be a 10/10 match, a 9/10 match, or an 8/10 match if one of the mismatches is at DQB1.
* Related donor mismatched at one to five HLA alleles (haploidentical)
* Matched related donor may be considered suitable donors for this protocol if a peripheral stem cell donation is deemed by the clinical team to be a safer donation option (if donor is not a suitable candidate for a bone marrow harvest) or if there is concern that bone marrow harvest would not yield adequate cell doses Additionally, a matched related donor would be considered suitable for this protocol if there are safety concerns regarding a patient receiving a standard T cell replete bone marrow transplant due to individualized GVHD risk or risk related to standard GVHD prevention medications.
* Donor suitable for mobilization of peripheral stem cells and apheresis and fulfills infectious disease criteria as per our institutional SOP, including HIV, HepB, HepC PCR negative.
* We assess donor eligibility as per our Allogenic Donor Evaluation for Eligibility standard operating procedure. These procedures apply for determining donor eligibility, including donor screening and testing for relevant communicable disease agents and diseases. Our donor collection program is FACT accredited.
* Related donors will be consented and enrolled under IRB approved research protocol for cell collection per IRB 04-004078 CHP 784 Clinical and Research Collection and Future Research Use of Bone Marrow, Stem Cells or T Cells.
* Unrelated donor identified through the National Marrow Donor Program (NMDP) and fulfills the NMDP criteria for donation. Unrelated donor willing and able to undergo mobilization of peripheral stem cells and apheresis.
* The donors selected for this IDE will either be unrelated donors identified through the National Marrow Donor Program (NMDP) or related donors. Regarding the unrelated donors, NMDP procedures for determining donor eligibility include donor screening and testing for relevant communicable disease agents and diseases

Exclusion criteria:

* Uncontrolled bacterial, viral, or fungal infections
* Fully HLA matched sibling donor (fully matched related donors including siblings may be included in special circumstances)
* Donor unable to donate peripheral stem cells
* Pregnant Females

Min Age: 1 Month | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tim Olson, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States